CLINICAL TRIAL: NCT01553006
Title: A Comparison of Cefditoren Pivoxil 10 mg/kg/Day and Cefditoren Pivoxil 20 mg/kg/Day in Treatment of Childhood With Acute Rhinosinusitis
Brief Title: Study of Cefditoren Pivoxil in Treatment of Childhood With Acute Rhinosinusitis
Acronym: RS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Orapan Poachanukoon, Associate Professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-PE-5-036/54
Record Dates: First submitted 2012-02-17; First posted 2012-03-13 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Rhinosinusitis
Keywords: rhinosinusitis; cefditoren pivoxil
MeSH Terms: conditions — Rhinosinusitis | interventions — cefditoren pivoxil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cefditoren pivoxil (Active Comparator): cefditoren 10 mg/kg/day for 14 days
  Interventions: Drug: cefditoren pivoxil
- cefditoren pivoxil high dose (Active Comparator): cefditoren 20 MKD were used to compare efficacy of treatment.
  Interventions: Drug: cefditoren pivoxil

INTERVENTIONS:
Drug: cefditoren pivoxil — comparison of different dosages of cefditoren pivoxil
  Other Names: Meiact

SUMMARY:
Cefditoren pivoxil has been used in rhinosinusitis treatment. However, little is known about the efficacy of this drug at low and high doses.

DETAILED DESCRIPTION:
The investigation was a randomized, investigator-blinded, and parallel study, conducted in patients (age 1-15 years) with acute rhinosinusitis. Two groups of patients were randomized received low (10 MKD) or high (20 MKD) of drug for 14 days. Changes in sinus symptoms scores, response rate and adverse effect were evaluated at days 7 and 14. Relapse rate was recorded at days 21 and 28. Recurrence of sinus symptoms at day 60 were assessed.

ELIGIBILITY:
Inclusion Criteria:

* children age 1-15 years old diagnosed acute rhinosinusitis

Exclusion Criteria:

* poor compliance
* other infections

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
sinus symptoms scores | 14 days
  Change of sinus sympotms scores from baseline in 2 weeks

SECONDARY OUTCOMES:
relapse rate | at day 28
  The relapse rate of sinus symptoms scores at day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Orapan Poachanukoon, MD., Principal Investigator — Thammasat University
Locations (1):
- Thammasat University, Prathumthani, Thailand